CLINICAL TRIAL: NCT03833323
Title: Implantable System for Remodulin Post-Approval Study
Acronym: ISR PAS
Status: Withdrawn | Type: Observational
Why Stopped: Implantable System for Remodulin not commercially approved.
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Collaborators: United Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: ISR PAS
Record Dates: First submitted 2019-02-05; First posted 2019-02-07 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: PAH; Pulmonary Arterial Hypertension; Pulmonary Hypertension; Remodulin; treprostinil; DelIVery for PAH; Implantable Pump; Drug Pump; Intrathecal Catheter; Targeted Drug Delivery; Programmable Pump
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hypertension, Pulmonary | interventions — treprostinil

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Combination Product: Implantable System for Remodulin (treprostinil) — All patients will be implanted with the Implantable System for Remodulin (treprostinil).

SUMMARY:
The purpose of the Implantable System for Remodulin (ISR) Post Approval Study (PAS) is to provide evaluation and periodic reporting of the safety and effectiveness of Medtronic market-released ISR, including the catheter and the pump.

DETAILED DESCRIPTION:
The ISR PAS is an observational, prospective, non-randomized, multi-center study. It will enroll a minimum of 50 newly implanted patients at up to 10 US sites, observing and reporting catheter-related complications and pump failures through 5 years post implant.

ELIGIBILITY:
Inclusion Criteria:

* Subject or legally authorized representative provides written authorization and/or consent per institution and geographical requirements.
* Subject is intended to receive an eligible ISR product.
* Subject is at least 22 years of age.

Exclusion Criteria:

* Subject is pregnant.
* Subject who is expected to be inaccessible for follow-up.
* Subject with exclusion criteria required by local law.
* Subject is currently enrolled in or plans to enroll in any concurrent drug and/or device study that may confound results (i.e. no required intervention that could affect interpretation of all-around product safety and or effectiveness).

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly implanted patients that are intended to receive an ISR.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Catheter-related complications | Implant to 5 years post-implant
  Number of adverse events requiring invasive intervention that are related to the ISR catheter.
Pump failures | Implant to 5 years post-implant
  Number of adverse events requiring invasive intervention that are related to the ISR pump.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bourge, MD, Study Chair — University of Alabama at Birmingham